CLINICAL TRIAL: NCT03058471
Title: Efficacy of Starting Methotrexate Early in Chikungunya Arthritis:A 24 Week Randomized Controlled Open Label Crossover Trial
Brief Title: Efficacy of Starting Methotrexate Early in Chikungunya Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Shefali khanna sharma, Assosciate professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NK/3088/STUDY
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Early Chikungunya Arthritis
MeSH Terms: interventions — Methotrexate; Anti-Inflammatory Agents, Non-Steroidal; Steroids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- methotrexate (Active Comparator): mehotrexate 10 mg weekly, to be increased by 5 mg in each visit to a maximum of 25 mg
  Interventions: Drug: Methotrexate; Drug: Steroids
- non steroidal anti inflammatory drugs (Active Comparator): NSAID in full dose with Pantoprazole. If remission not achieved at 2 months, will be given methotrexate as in methotrexate arm
  Interventions: Drug: NSAID; Drug: Steroids

INTERVENTIONS:
Drug: Methotrexate — methotrexate arm will be given methotrexate starting at 10 mg weekly to be increased to 25 mg maximum in subsequent visits gradually
  Arms: methotrexate
Drug: NSAID — this arm will be given NSAID to the tolerable full dose with pantoprazole
  Arms: non steroidal anti inflammatory drugs
Drug: Steroids — inj. depot methyl prednisolone 80 mg ,2 doses deep intramuscularly given one week apart to all patients who have 5 or more swollen or tender joints

SUMMARY:
This is a single center, prospective, randomized controlled open label trial with a one sided cross over design to compare the efficacy of initiating Methotrexate(Mtx) in early post Chikungunya induced arthritis (4-12 weeks after onset) with Non Steroidal Anti inflammatory Drugs(NSAID) alone.

DETAILED DESCRIPTION:
This will be a single center, prospective, randomized controlled open label trial with a cross over design. Patients will be recruited from outpatient department of internal medicine and rheumatology clinic of Post Graduate Institute of Medical Education and Research(PGIMER), Chandigarh, India, a tertiary care hospital. .

Inclusion Criteria

1. Patients of confirmed Chikungunya virus infection as per World Health Organisation(WHO) guidelines defined as atleast one of the following

   1. Presence of viral ribonucleic acid in sera determined with Real Time Polymerase Chain Reaction(RT PCR) in acute phase < 7 days of fever
   2. Presence of virus specific IgM antibodies in serum
2. Persistent arthritis after 4 weeks of onset of fever and duration less than 12 weeks(early post viral arthritis)
3. Age more than 16 years
4. Patients willing to give informed consent

Exclusion Criteria:

1. Patients with mixed infection i.e. dengue.
2. Having a known rheumatological disease and currently taking treatment
3. Pregnant and breastfeeding women
4. Any contraindication to methotrexate(Mtx)

The clinical details of patients will be recorded in the proforma which includes details regarding the fever and musculoskeletal symptoms.

At baseline, a complete blood count (CBC), erythrocyte sedimentation rate (ESR), C-Reactive protein(CRP), liver function tests(LFT), Renal Function Test(RFT), rheumatoid factor (RF), anti- citrullinated peptide antibodies (ACPA) will be done. All eligible patients will be randomized to two groups. Randomization will be done by computer generated block randomization in blocks of four and six. In one group methotrexate will be started at a dose of 10 mg/week after checking basal CBC,LFT and RFT and will be increased gradually(5mg/each visit)to 25 mg if there is no response at subsequent visits and the other group will be continued on NSAID.If remission (no swollen or tender joints at the visit) is not achieved in the NSAID group at 2 months they will be given MTX .MTX group will be given NSAID on need basis and this will be recorded in each visit. Both groups will be given depot methyl prednisolone 80 mg ,2 doses 1 week apart if there is 5 or more swollen or tender joints at any visit.The patients will be assessed at 0,1, 2,4 and 6 months for Tender Joint Count(TJC),Swollen joint count( SJC) and Indian Health Assessment Questionnaire(HAQ). If a patient achieves remission in methotrexate group, the last dose of methotrexate will be continued till next visit. The dose will be halved in the next visit and stopped in the next.In the NSAID group, if remission is achieved, dose will be changed to on need basis and if the patient relapses will be started on methotrexate. Allocation concealment will be ensured by means of enclosing the randomization sequence in sealed opaque envelopes. One of the investigator, blinded for the treatment received by the subjects, will assess the subjects at recruitment to the study and subsequently during their next visits and at the end of study period.

Primary efficacy end point will be proportion of patients achieving remission (No tender or swollen joint)at 6 months. Secondary end points will be the time duration to achieve remission, change in DAS28 ESR/CRP score, proportion of patients achieving remission by simplified disease activity index(SDAI) and clinical disease activity index( CDAI) score, functional status assessed by Health Assessment Questionnaire-Indian version (HAQ) , change in pain VAS(Visual Analogue Scale) 100mm,adverse effects and the difference in NSAID and intra muscular steroid injection requirement among the groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of confirmed CHIK-V infection as per WHO guidelines defined as atleast one of the following

   1. Presence of viral ribonucleic acid in sera determined with RT -PCR in acute phase < 7 days of fever
   2. Presence of virus specific IgM antibodies in serum
2. Persistent arthritis after 4 weeks of onset of fever and duration less than 12 weeks
3. Age more than 16 years
4. Patients willing to give informed consent

Exclusion Criteria:

1. Patients with mixed infection i.e. dengue.
2. Having a known rheumatological disease and currently taking treatment
3. Pregnant and breastfeeding women
4. Any contraindication to methotrexate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
remission | 6 months
  no swollen or tender joints

SECONDARY OUTCOMES:
change in DAS 28 ESR/CRP | at 6 months
change in functional status assessed by Health Assessment Questionnaire-Indian version (HAQ) | at 6 months
time to remission | at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes
all study data can be available after the study completion. Contact the auther.